CLINICAL TRIAL: NCT03206307
Title: Spiroergometrische Und Psychologische Messungen Zur Vorhersage Der Erwerbsfähigkeit Und Rückkehr Zur Arbeit Nach 18 Und 36 Monaten Nach Der Medizinischen Rehabilitation
Brief Title: Spiroergometric and Psychological Measurements to Predict Return to Work After 18 and 36 Months After Medical Rehab
Acronym: SPIRO
Status: Completed | Type: Observational
Sponsor: Jacobs University Bremen gGmbH (Other)
Responsible Party: Sponsor
Other Study IDs: 060.001.12.00 - 3.050
Record Dates: First submitted 2017-06-08; First posted 2017-07-02 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Employability
Keywords: Return to work; medical rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group 1 will be questioned 36 months (in 2017) after their medical rehabilitation which was in 2013/2014.
- Group 2: Group 2 has the medical rehabilitation in 2017 and will be questioned at the end of the medical rehabilitation and 6, 12 and 18 months after that

SUMMARY:
Can professional performance and the probability of returning to work up to three years after medical rehabilitation be predicted by spiroergometric data (or performance of the cardiovascular system) together with psychological factors (motivation, self-efficacy) as well as physical activity, and their interaction? How are work related and health related factors associated with the The following variables: workload, work satisfaction, personal assessment of the professional future and psychological stress?

DETAILED DESCRIPTION:
One main aim of medical rehabilitation is to restore ability to work. The goal is to increase health, as well as the performance and functional capacity of the the rehabilitant, in order to improve their occupational ability, as well as social activity and participation.

A number of the psychological and structural factors involved in this are already known. There is less evidence, however, regarding the importance of objectively measured performance and functioning, as well as the relation of these objective measures with subjective factors (i.e., the interaction of cardiovascular performance and physical activity with psychological factors with).

Therefore, this study investigates how rehabilitants can successfully decrease their professional vulnerability, and the importance of spiroergometric and psychological data to predict viability and return to work.

The aim is to improve the theorised variance in predicting the viability and return to work and, based on the results, to make appropriate recommendations to those affected and their social network, rehabilitation facilities, those offering rehabilitation services, employers and physicians.

The following research questions are to be answered with this study:

1. Can spiroergometric data and psychological mechanisms characterize:

   (A) workability and physical activity, (B) self assessment of the professional future, (C) return to working life, (D) ability to deal with occupational burdens (professional capacity)

   ... 6, 12, 18 and 36 months after medical rehabilitation?
2. What is the significance of objective data compared to subjective characteristics (such as "higher level goals" in terms of employment), and how are the mediating psychological mechanisms involved?

In rehabilitation patients with degenerative skeletal diseases, a spiroergometry measurement (cardiovascular checkup) was carried out in 2013/2014 (group 1, G1). This study determined the performance of the cardiovascular system and the general "fitness". The patients were also questioned about age, workload, work satisfaction, assessment of the future of the profession and accompanying psychological stress.

A follow-up survey of those who are insured is to be carried out by telephone.

In addition, new patients (group 2, G2) are to be interviewed and spiroergometrically tested, as well as to be interviewed three times over the phone.

This will allow: (1) analyzing the change over time and the cardiovascular capacity beyond psychological factors (motivation, self-efficacy) and physical activity, (2) comparisons with other insured persons.

Data collection after rehabilitation is carried out as a computer-assisted telephone interview, and is conducted after the rehabilitation after 6, 12, 18 (G2) and 36 months (G1).

ELIGIBILITY:
Inclusion Criteria:

* Degenerative skeletal disease
* Medical rehabilitation at Montanus-Klinik Bad Schwalbach
* Insured with the Deutsche Rentenversicherung Oldenburg-Bremen
* Sufficient knowledge of the German language
* Telephone or mobile phone connection

Exclusion Criteria:

* Insufficient knowledge of the German language
* No participation in the spiroergometrical measurement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the study insured members of the Deutsche Rentenversicherung Oldenburg-Bremen with a granted medical rehabilitation treatment at the Montanus-Klinik Bad Schwalbach will be asked to fill out a questionnaire when arriving at the rehabilitation clinic as well as to take part in three subsequent telephone interviews after 6,12 and 18 months.
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Oxygen absorption during stress test | 6 months
  Measured by VO2MAX (maximum oxygen consumption in ml / kg body weight / min)
Workability, as measured by questionnaire - change at 6, 12 and 18 months + at 36 months after rehabilitation | After the rehabilitation treatment at 6, 12 and 18 months (G2) + at 36 months (G1)
  Parameters include health status, employment history, current position, working hours, physical, mental or emotional restrictions to work
Job satisfaction, as measured by questionnaire - change at 6, 12 and 18 months + at 36 months after rehabilitation | After the rehabilitation treatment at 6, 12 and 18 months (G2) + at 36 months (G1)
  Parameters include earning capacity, whether job is mentally/physically/emotionally/inter-personally exhausting, skills required, whether recognition is received, independence, boring/challenging , overwhelming, continuous learning, whether important to the person
Personal appraisal of the professional future, as measured by questionnaire - change at 6, 12 and 18 months + at 36 months after rehabilitation | After the rehabilitation treatment at 6, 12 and 18 months (G2) + at 36 months (G1)
  Parameters include whether individual expects future work difficulties professionally and/or due to health restrictions
Return to working life, as measured by questionnaire - change at 6, 12 and 18 months + at 36 months after rehabilitation | After the rehabilitation treatment at 6, 12 and 18 months (G2) + at 36 months (G1)
  Parameters include how many hours individual desires to work again
The handling of occupational burdens, as measured by questionnaire - change at 6, 12 and 18 months + at 36 months after rehabilitation | After the rehabilitation treatment at 6, 12 and 18 months (G2) + at 36 months (G1)
  Parameters include personal initiatives to make return to work practical: changing working conditions, reduction in work hours, different position, professional training, attended health promoting courses, attended coaching/counseling, engaged in self-help, lifestyle changes

SECONDARY OUTCOMES:
Plans to participate and wishes to take measures to safeguard the earning capacity, as measured by questionnaire - change at 6, 12 and 18 months + at 36 months after rehabilitation | After the rehabilitation treatment at 6, 12 and 18 months (G2) + at 36 months (G1)
  Parameters include personal reasons to safeguard earning capacity: money, feeling needed, interpersonal contact, recognition, knowledge/experience, fun, routine, development, mentally fitness, being outside the home, purpose in life, expectations from others, physical fitness, distraction from other problems
Self-imposed objectives and achievement, as measured by questionnaire - change at 6, 12 and 18 months + at 36 months after rehabilitation | After the rehabilitation treatment at 6, 12 and 18 months (G2) + at 36 months (G1)
  Parameters include personal objectives to achieve from rehabilitation: improved mobility, improved physical condition, improved physical illness and complaints, improved mental condition, improved interpersonal situation, improved professional situation, improved working capacity, weight loss, pain reduction, overall health promotion, deal with daily stress, more confidence
Personal, social and contextual factors, as measured by questionnaire - change at 6, 12 and 18 months + at 36 months after rehabilitation | After the rehabilitation treatment at 6, 12 and 18 months (G2) + at 36 months (G1)
  Parameters include: perceived job security, earning capacity risk, satisfaction with life, satisfaction with job-related activities, satisfaction with physical activity, social support, self-efficacy
Participation in interventions, as measured by questionnaire - change at 6, 12 and 18 months + at 36 months after rehabilitation | After the rehabilitation treatment at 6, 12 and 18 months (G2) + at 36 months (G1)
  Parameters include participation in: medical treatments, psychological therapies, disease-specific group training, physical therapy, movement therapy, general health training, work-related measures, professional advice, relaxation techniques

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Prof. Dr., Principal Investigator — Jacobs University Bremen gGmbH
Locations (1):
- Jacobs University Bremen gGmbH, Bremen, Germany

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan.

REFERENCES:
- [Derived] Rinn R, Gan Y, Whittal A, Lippke S. Cardiopulmonary capacity and psychological factors are related to return to work in orthopedic rehabilitation patients. J Health Psychol. 2021 Nov;26(13):2505-2519. doi: 10.1177/1359105320913946. Epub 2020 Apr 28. PMID 32345071